CLINICAL TRIAL: NCT03195985
Title: Managing Stress and Cognitive Difficulties With a Short Mindfulness-based Intervention in Old Adults With Subjective Cognitive Complaints
Brief Title: Mindfulness in Old Adults With Subjective Cognitive Complaints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: University of Westminster (Other); Imperial College London (Other)
Responsible Party: Principal Investigator, Marcela P. Vizcaychipi, Consultant in Anaesthesia and Intensive Care, Chelsea and Westminster NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C&W1234
Record Dates: First submitted 2016-12-02; First posted 2017-06-22 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Subjective Cognitive Complaints; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Intervention (Experimental): Mindfulness intervention of 4 weeks
  Interventions: Other: Mindfulness-based intervention
- "Age Well" psycho-education course (Active Comparator): 4-week active control condition
  Interventions: Other: Age Well psycho-education

INTERVENTIONS:
Other: Mindfulness-based intervention — A shortened, 4 week mindfulness intervention course based on the original 8 week mindfulness-based stress reduction course by Jon Kabat-Zinn
  Arms: Mindfulness-based Intervention
Other: Age Well psycho-education — 4-week active control condition aimed at psycho-education regarding healthy ageing
  Arms: "Age Well" psycho-education course

SUMMARY:
The study will focus on measuring stress, rumination and cognitive function across three time points in old adults with subjective cognitive complaints via a 4-week short mindfulness intervention, as compare to an active control condition (psycho-education course "ge Well").

This is a pilot study.

DETAILED DESCRIPTION:
20 old adults with subjective cognitive complaints will be recruited from adult day centres and the Chelsea Westminster Hospital in London. All patients will be aged 65 and above. Each participant will be randomly allocated to either a mindfulness intervention or the active control condition (psychoeducation) with 10 participants in each intervention.

A short mindfulness intervention of 4 weeks will be delivered by a trained mindfulness teacher across four 2 hour sessions that focus on the breath, links between mind and body, sensory and metacognitive awareness, emotion regulation, movement and compassion using visually engaging materials that will enhance understanding, encoding and recollection.

There will be one session per week. The proposed study will evaluate the effects of a short mindfulness intervention in old adults with subjective cognitive complaints. Management of emotional difficulties associated with anxiety and stress can improve psychological well-being in sufferers, and in turn can enhance cognitive capacity to maximise function. Mindfulness interventions are gentle, non-invasive and cost effective techniques that have been designed for stress reduction, that have been associated with improvements in mood, stress, pain management and overall well-being in a range of clinical and healthy populations. In addition mindfulness interventions have also been shown to improve cognitive function and emotion regulation by enhancing attentional awareness, attentional flexibility and attentional capacity. However, very few studies to date focus on elderly participants and no study to date has tried to shorten the current 8-week Mindfulness-Based Stress Reduction training in older adult populations.

The psycho-education course will also take 4 consecutive weeks, with one session each week.

All participants will be screened (see Appendix 6 of protocol) prior to the beginning of the study and recruited if they fulfil the criteria required as highlighted within the 'participants' section. The screening session will take approximately 20minutes. Written informed consent will be obtained from the participant prior to performing any study related evaluations or procedures. Informed consent (see Appendix 4 of protocol) will be taken during all assessment sessions and also during the screening assessment.

Participants will be provided with written information about the study in the form of a participant information sheet (see Appendix 3 of protocol) and mindfulness course leaflet, and will be allowed a minimum of 24 hours for questions and to consider the study before agreeing to participate. It will be the responsibility of the investigator or co-investigator to obtain written informed consent prior to undertaking any questionnaires, tests, or hair sampling detailed within the protocol.

The Mini-Mental State Examination and the National Adult Reading Task will be performed during a screening session only. All other assessments (cognitive, psychological and physiological) will be done at baseline, pre- intervention (week 4), and at a follow-up (week 8).

All assessments done during baseline, week 4, and week 8 assessment sessions will take approximately 45minutes per session. Each assessment session will follow the same order in which questionnaires and tasks are presented to participant (see Appendix 5 of protocol).

Physiological assessment: Hair cortisol will be sampled from each participant during the three assessment stages (baseline, week 4, and 8) by obtaining hair samples from participant's vertex posterior. Each sample will be approximately 0.5cm in diameter, and will be used for analysis carried out by Stratech (formerly Salimetrics) whereby 10% of the sample will be extracted in duplicate and the remaining 90% of extractions will be performed in singlet. Individually wrapped hair samples will be stored at a temperature between 20 and 25 degrees Celsius in a breathable container. The sampling should take approximately 5 minutes for each participant.

The following hair sampling equipment is not included by Stratech and will need to be provided by the researcher: thread for tying hair samples, sharp scissors, hair clips, a pin-tailed comb, aluminium foil, large paper envelopes for long-term storage, and jiffy bags for shipping.

Cognitive Assessment: The cognitive domain will be assessed based on the Trail Making Task (TMT) at three time points (baseline, week 4, and 8) and will provide information on executive function, and also based on the Verbal Fluency Tasks to assess verbal fluency and executive function. The Everyday Memory Questionnaire (EMQ) will be used to assess subjective memory function at the three time points (baseline, week 4, and 8). The Verbal Fluency Tasks will consist of the FAS phonemic fluency task and the Animal Naming Task (semantic fluency).

Psychological Assessment: The psychological domain will be assessed based on the Perceived Stress Scale (PSS) which will provide information on the subjective stress levels of participants, and also based on the Penn State Worry Questionnaire - Abbreviated (PSWQ-A) which will provide information on the amount of worry each participant feels, and also the Rumination Response Scale (RRS) which will provide information regarding the effect of mindful exercises on ruminative behaviours. These will all be assessed at the three assessment points (baseline, week 4, and 8).

Please note all questionnaires and tasks involved are validated.

All questionnaires and tasks will be administered in paper form in the presence of a member of the research team trained at administering the tasks.

The Mindfulness course:

A short mindfulness course will be delivered by a trained mindfulness teacher and Clinical Psychologist across four 2-hour sessions.

The course will be accompanied by a booklet designed by Edginton and Nenadlova (in prep) highlighting the main themes within each session using visually engaging pictures to help enhance understanding, encoding and recollection (see appendix 1 of protocol).

There will be one session per week for 4 consecutive weeks, at the same time each week. The details of each session are described below:

Week 1:

Introduction to the topic. Guided mindful eating. Focus on being 'in the moment' and appreciating the task the participant doing at each point in time.

Mindful eating will take form via eating a raisin - studying the raisin in detail (colour, sensations such as smell and texture) and focusing in detail on the process involved in eating the raisin.

The aim of this session will be to teach participants to focus on each task that they are doing in detail, with the goal to be able to give full attention to each task, without thinking about the next task.

Homework given in the form of a practice exercise.

Week 2:

Recap of the previous week's topic. Guided mindful breathing exercise, focus on the breath and being 'in the moment'.

Guided mindful body-scan. Focus on different parts of the body and its sensations via a guided body scan exercise.

Emphasis on observing sensations rather than judging sensations. Focus on being 'in the moment', focusing at one thing at a time, and also training the ability to focus attention and awareness to different parts of the body at will.

Homework given in the form of a practice exercise.

Week 3:

Recap of the previous week's topic. Guided session mindful coping and dealing with difficulties. The aim of the session will be to become mindfully aware of whatever is most predominant in the participant's moment by moment experience, and for participants to uncover how they are relating to feelings and thoughts are arising, and approach them in an accepting way.

Exercise practiced during the session: The Three Step Breathing Space - creating an imaginary space around ourselves by imaging our breath expanding beyond our body into the space around us.

Homework given in the form of a practice exercise.

Week 4:

Recap of the previous week's topic. Guided session on mindful choices and looking after own self. Exercises involve (a) focusing on what the participant finds nourishing and depleting in their daily activities and (b) a guided Mountain exercise whereby participants imagine themselves as being a mountain which stands tall despite the ever-changing environment around them. Recap of topics covered will be included at the end, and suggestion for how to continue the practice beyond the course will be provided.

The delivery of the mindfulness intervention will be designed for independent groups of up to 10 participants within one class.

The active control condition:

The active control condition will be identical in length to the mindfulness course. It will consist of 4 "Age Well" psycho-education sessions. These sessions will aim to provide individuals with knowledge about general well-being such as healthy movement and activity, healthy eating, and the importance of cognitive stimulation.

These sessions will run in parallel to the mindfulness course, and will be run by the Clinical Psychologist.

Participants will be asked to write their name onto an attendance sheet during both Mindfulness and "Age Well" sessions to track participant attendance throughout the courses (Appendix 2 of protocol).

Please note that the screening and assessment visits may take place within +/- 7 days based on the discretion of the Chief Investigator. Date of each assessment visit will be recorded on the informed consent form which will be signed at each assessment visit.

The research is being funded by the Imperial College Alzheimer's Network, London.

ELIGIBILITY:
Inclusion Criteria:

* All willing and consenting patients over the age of 65
* Patients who have been admitted to the hospital and who have been formally diagnosed with MCI at the Memory Clinic
* Patients with hair at the posterior vertex
* Patients with fluent English
* Patients who can commit to the entire length of the study
* Patients with interest in mindfulness

Exclusion criteria:

* Being under 65 years of age
* Presence of any psychiatric disorders,
* Presence of myopathy
* Presence of atherosclerosis
* Use of steroids
* Having undergone chemotherapy
* heart disorder
* dementia
* head injury
* advanced neurodegenerative disease
* any patient having had dyed their hair less than one week prior to the first cortisol sampling

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in cortisol levels between the two MCI groups over time | One month
  assessed by collecting hair from the vertex posterior for stress hormone analysis

SECONDARY OUTCOMES:
Changes in anxiety over time | One month
  Beck's Anxiety Inventory
Changes in verbal learning and memory over time | One month
  Mini-Mental State Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Trudi Edginton, PhD, Principal Investigator — Chelsea & Westminster Hospital, London UK
Locations (2):
- United Kingdom (2):
  - Chelsea and Westminster Hospital NHS Trust, London
  - The Magill Department of Anaesthesia, Chelsea and Westminster Hospital, London

IPD SHARING:
Plan to Share IPD: No